CLINICAL TRIAL: NCT01105117
Title: An Open-label Extension of Study AC-066A401 Investigating the Safety and Tolerability of ACT-385781A Compared to Flolan® in Injectable Prostanoid Treatment-naïve Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Epoprostenol for Injection in Pulmonary Arterial Hypertension - Extension of AC-066A401
Acronym: EPITOME-1 Ext
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-066A402
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; EPITOME-1
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ACT-385781A (Actelion Epoprostenol)
  Interventions: Drug: ACT-385781A (Actelion Epoprostenol)
- 2 (Active Comparator): Flolan®
  Interventions: Drug: Flolan®

INTERVENTIONS:
Drug: ACT-385781A (Actelion Epoprostenol) — per Prescribing Information
  Arms: 1
Drug: Flolan® — per Prescribing Information
  Arms: 2

SUMMARY:
This is an open-label, non-randomized extension to study AC-066A401. The study will assess safety and tolerability of ACT-385781A and Flolan (epoprostenol sodium) while providing a means for continuing treatment after ending participation in study AC-0066A401.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-mandated procedure
2. Patients who completed participation in study AC-066A401
3. Patients who have not obtained authorization for commercial ACT-385781 and Flolan at the time of ending participation in study AC-066A401

Exclusion Criteria:

1. Patients who prematurely discontinued study drug in study AC-066A401
2. Patients for whom continued treatment with either ACT-385781 and Flolan is no longer considered appropriate
3. Known hypersensitivity to the investigational drug or comparative drug or drugs of the same class, or any of their excipients
4. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease
5. Known concomitant life-threatening disease with a life expectancy < 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Benton, PharmD, Study Director — Actelion
Locations (7):
- United States (7):
  - University of California - San Diego, La Jolla, California
  - University of Colorado - Denver, Aurora, Colorado
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania-Penn Presybyterian Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at Pulmonary Hypertension centers in the U.S.
Pre-assignment Details: In this extension study patients could continue on the randomized treatment they received in the core study (AC-066A401) until commercial treatment became available.
Groups:
- ACT-385781A (Epoprostenol for Injection): ACT-385781A (Actelion Epoprostenol)
  ACT-385781A (Actelion Epoprostenol) : per Prescribing Information
- Flolan® (Epoprostenol Sodium) for Injection: Flolan®
  Flolan® : per Prescribing Information
Period: Overall Study
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (0) | 34 (0) | 44.5 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of ACT-385781A and Flolan in Injectable Prostanoid Treatment-naïve Patients With Pulmonary Arterial Hypertension (PAH) - Number of Patients With Adverse Events Leading Discontinuation of Study Treatment
Time Frame: Up to 39 days. Day 1 - until patients transition from study medication to commercially-obtained medication
Population: Study population
Measure: Number; unit: participants
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

2. Primary Outcome: Safety and Tolerability of ACT-385781A and Flolan in Injectable Prostanoid Treatment-naïve Patients With PAH - Number of Deaths
Time Frame: Up to 39 days. Day 1 - until patients transition from study medication to commercially-obtained medication
Population: Study population
Measure: Number; unit: participants
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening to day 28 for treatment-emergent (TE) adverse events (AEs) up to day 28 (EOT). TE serious AEs (SAEs) up to 30 days post study drug.
Description: Assessment of safety was based on the collection of AEs, including SAEs and AEs that resulted in discontinuation of study treatment. All AEs that occurred up to the end of the last day of study treatment were recorded in the CRF and included in the clinical database. SAEs and deaths that occurred up to 30 days after the end of study treatment.
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACT-385781A (Epoprostenol for Injection) (N=1) | Flolan® (Epoprostenol Sodium) for Injection (N=1)
Right ventricular failure (Cardiac disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACT-385781A (Epoprostenol for Injection) (N=1) | Flolan® (Epoprostenol Sodium) for Injection (N=1)
Catheter site erythema (General disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No